CLINICAL TRIAL: NCT00055484
Title: A Double-Blind, Randomized, Multicenter, Parallel Dose Study to Evaluate the Safety and Efficacy of Zonisamide 150 mg and 300 mg Per Day and Placebo in Subjects With Migraine Headache
Brief Title: A Study to Measure the Safety and Effectiveness of Zonisamide in Subjects With Migraine Headache
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elan Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AN46046-228
Record Dates: First submitted 2003-03-03; First posted 2003-03-05 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Migraine Headache
Keywords: Migraine Headache; prophylaxis; AED; migraine prophylaxis
MeSH Terms: conditions — Migraine Disorders | interventions — Zonisamide

INTERVENTIONS:
Drug: zonisamide

SUMMARY:
The purpose of this study is to determine if zonisamide is effective as a preventative medication for individuals with migraine headache.

DETAILED DESCRIPTION:
The pharmacologic treatment of migraine may be acute (abortive, symptomatic) or preventive (prophylactic). Preventive medication is usually given daily for months or years; however, treatment may also be given in an intermittent regimen. Most migraine prophylactic medications were designed to treat other disorders, and they can be divided into three groups:

1. Serotonergic or monoaminergic agents such as methysergide, which have demonstrated high degrees of effectiveness;
2. Non-serotonergic drugs such as beta-blockers, tricyclic antidepressants, valproate; and
3. Drugs with lesser demonstrated effectiveness, such as selective serotonin reuptake inhibitors, calcium channel antagonists, and non-steroidal anti-inflammatory drugs.

The choice of treatment must be individualized, and is influenced by contraindications, potential side effects, the need to treat associated symptoms like tension-type headache and insomnia, and drug cost.

Anticonvulsants, such as valproate, have shown significant degrees of efficacy in migraine prophylaxis when used in low doses. Considering the differences in proposed mechanisms of action of these agents, it is likely that a novel anticonvulsant such as zonisamide may also be an effective prophylactic treatment for migraine.

ELIGIBILITY:
INCLUSION:

Subjects who meet all the following criteria will be eligible to participate in the study:

* Are men or women, between the ages of 18 and 65, inclusive.
* Satisfy diagnostic criteria for migraine headache, consistent with criteria described in Headache Classification Criteria.
* Have at least 4 migraine attacks per 28 days [each attack separated by at least 48 hours] prior to the Screening Visit and experience at least 4 migraine attacks during the Screen/Baseline Phase.
* Agree to not become pregnant during the study and agree to use an adequate method of birth control during the study such as an adequate barrier method, hormonal contraceptive, or surgical sterilization. All women of childbearing potential must have a negative pregnancy test before entering the study and during the study.
* Are able to swallow the capsules whole.
* Are willing and able to follow Investigator instructions and study procedures, complete the daily diary, and report adverse events.

EXCLUSION:

Subjects meeting any of the following criteria will not be eligible to participate in this study:

* Have required more than 3 different rescue medications for control of a single attack anytime within 3 months prior to the Screening Visit.
* Have cluster headache or chronic tension type headache and are unable to distinguish between their different types of headache.
* Have basilar or hemiplegic migraine.
* Have used triptans more than 3 times per week within 3 months prior to the Screening Visit.
* Have received botulinum toxin injection(s) within 3 months prior to the Screening Visit.
* Have taken any other prophylactic medications for migraine within 5 half-lives prior to the Baseline Visit.
* Are pregnant or lactating.
* Have a history or current diagnosis of psychiatric disorder likely to require pharmacological intervention (e.g., antidepressants, MAO inhibitors, antipsychotics, mood-stabilizers, anxiolytics) during the study.
* Have clinically unstable cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease.
* Have laboratory test results that, in the opinion of the Investigator, are clinically significant abnormalities.
* Require treatment with any medication (e.g., daily opioids, daily beta-blockers, daily non-steroidal anti-inflammatory drugs, carbonic anhydrase inhibitors, eletriptan) or herbal supplements (e.g., St. John's Wort, ginseng, ginkgo biloba, kava kava, melatonin, petadolex) that might interact adversely with, or obscure, the action of the study medication.
* Have received psychoactive medication (e.g., other anticonvulsant drugs, antidepressants, antipsychotics, anxiolytics, mood stabilizers) within 5 half-lives prior to the Baseline Visit.
* Have previously enrolled in this study or previously treated with zonisamide.
* Have previously failed an adequate trial of another antiepilepsy drug for the treatment of migraine.
* Have a history of allergy or hypersensitivity to zonisamide or other sulfonamides.
* Have a history of skin rash, without other diagnosis, associated with any medication or any medical condition.
* Have a history of nephrolithiasis.
* Have received an experimental drug or used an experimental device within 30 days of the Screening Visit.
* Have a history of drug or alcohol abuse within 12 months prior to the Screening Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204
Dates: Start 2002-03; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Medical Affiliated Research Center, Huntsville, Alabama
  - University of South Alabama Medical Ctr Department of Neurology, Mobile, Alabama
  - Valley Neurological Headache Clinic, Phoenix, Arizona
  - The New England Center for Headache, Stamford, Connecticut
  - Radiant Research, Overland Park, Kansas
  - Michigan Head-Pain & Neurological Institute, Ann Arbor, Michigan
  - Mercy Health Research, Chesterfield, Missouri
  - Headache Care Center, Springfield, Missouri
  - Neurological Associates of Tulsa, Tulsa, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - MetaClin Research, Austin, Texas
  - Houston Headache Clinic, Houston, Texas
  - Radiant Research, Salt Lake City, Utah